CLINICAL TRIAL: NCT03182166
Title: Pharmacokinetic and Pharmacodynamic Study of Golimumab in Ulcerative Colitis (UC) Patients With Loss of Response (LOR) Followed by Dose Optimization
Brief Title: Golimumab in Ulcerative Colitis (UC) Patients With Loss of Response (LOR) Followed by Dose Optimization
Acronym: GOLILOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1608162; 2016-004245-85 (EudraCT Number)
Record Dates: First submitted 2017-05-29; First posted 2017-06-09 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Ulcerative Colitis
Keywords: golimumab; clinical response; mayo score; rectosigmoidoscopy; ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — golimumab; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients treated with golimumab (Experimental): The optimization procedure is:
  * For patients treated at 50 mg of golimumab every 4 weeks (less than 80 kg) will have an increase dose of golimumab: 100 mg every 4 weeks for 8 weeks. They will have rectosigmoidoscopy for measured mayo score and blood samples for measured the concentration of golimumab antibodies.
  * For patients treated at 100 mg of golimumab every four weeks (more than 80 kg) will have an increase dose of golimumab: treated at 100 mg every 2 weeks for 4 weeks.
  They will have rectosigmoidoscopy for measured mayo score and blood samples for measured the concentration of golimumab antibodies.
  Interventions: Drug: Golimumab (Optimization); Diagnostic Test: Rectosigmoidoscopy; Biological: Blood samples

INTERVENTIONS:
Drug: Golimumab (Optimization) — Increase dose of golimumab.
  * For patients treated at 50 mg will be performed, dose will be intensified at 100 mg every four weeks.
  * For patients treated at 100 mg will be performed, dose will be intensified at 100 mg every two weeks while four weeks.
Diagnostic Test: Rectosigmoidoscopy — Rectosigmoidoscopy will be realized for calculated Mayo score
Biological: Blood samples — Blood samples will be collected for analysis the concentration of golimumab and antibodies to golimumab (ADAb) in the blood

SUMMARY:
It is planned to enroll 80 UC patients who will require optimization of golimumab after secondary LOR. The review of the study protocol and its approval by an Independent Ethics Committee of the University of Saint Etienne are pending. All patients enrolled will give their written informed consent before being included. This study will be conducted in accordance with the ethical principles that have their origins in the Declaration of Helsinki, in compliance with the approved protocol, good clinical practice and applicable regulatory requirements. Patients will visit the investigator from screening visit to visit 6 at W-1, W0, W2, W4, W8, and at the end of the follow-up at wk 24. During their participation, patients will record clinical parameters required to calculate the partial Mayo score reported over 3 days prior to the visit and endoscopy at W0, W2 (optional) , W4, W8 (optional) and at the end of the follow-up to calculate total Mayo score.

ELIGIBILITY:
Inclusion Criteria:

* Affiliate or beneficiary of social security
* Age>18 years
* Pregnant women or man
* Presenting primary response under golimumab induction and in loss of response during maintenance therapy
* Patient with an ulcerative colitis
* Treated with golimumab
* Signature of consent

Exclusion Criteria:

* Trying to become pregnant
* Mental or emotional disorders
* Patients with crohn's disease or indeterminate colitis
* cancer(<5)
* Patients not in agreement with this study protocol
* Patients with crohn's disease or indeterminate colitis
* Patients non primary responder to golimumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
correlation between concentration of golimumab and clinical response according to treatment | From baseline to 8 weeks
  Concentration of golimumab is measured by Enzyme Linked ImmunoSorbent Assay (ELISA).
  Clinical response is measured by the Mayo score.

SECONDARY OUTCOMES:
Number of patient with antibodies to golimumab | day 1
  Concentration of antibodies to golimumab is measured by Enzyme Linked ImmunoSorbent Assay( ELISA)
correlation between concentration of antibodies to golimumab and clinical response according to treatment | From baseline to 8 weeks
  Concentration of antibodies to golimumab is measured by Enzyme Linked ImmunoSorbent Assay (ELISA) Clinical response is measured by the Mayo score.
Number of patients with Infectious diseases or Neuropathies or Injection site pain or fever | up to 8 weeks
  Number of patients with Infectious diseases or Neuropathies or Injection site pain or fever

CONTACTS AND LOCATIONS:
Overall Officials: Xavier ROBLIN, MD PhD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (5):
- France (5):
  - CHU Amiens-Picardie, Amiens
  - CHU Lyon Sud, Lyon
  - CHU Montpellier - St Eloi, Montpellier
  - CHU Nice, Nice
  - Chu Saint Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No